CLINICAL TRIAL: NCT05093582
Title: The Headache-inducing Effects of Levcromakalim in Patients With Cluster Headache
Brief Title: The Effects of Levcromakalim in Patients With Cluster Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Professor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H20082689
Record Dates: First submitted 2021-09-17; First posted 2021-10-26 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Cromakalim; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator): Intravenous infusion of levcromakalim (1 mg/20 ml). The infusion is administered at constant speed by an automatic pump, lasting 20 minutes.
  Interventions: Drug: Levcromakalim
- Placebo (Placebo Comparator): Intravenous infusion of placebo (sterile saline, 20 ml). The infusion is administered at constant speed by an automatic pump, lasting 20 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — 12 active episodic patients, 15 episodic patients in remission and 20 chronic patients of both genders are randomized to receive a 20-minute infusion of levcromakalim and/or sterile saline on two days, with at least 3 days in between.
  Arms: Levcromakalim
Drug: Saline — 12 active episodic patients, 15 episodic patients in remission and 20 chronic patients of both genders are randomized to receive a 20-minute infusion of levcromakalim and/or sterile saline on two days, with at least 3 days in between.
  Other Names: Isotonic saline; 0.9% saline
  Arms: Placebo

SUMMARY:
Cluster headache is a primary headache disorder characterized by attacks of unilateral headache of short duration and severe pain intensity. There is an unmet need to understand the underlying disease mechanisms that will ultimately lead to the development of disease-specific medicines. Until now, it has been suggested that the calcitonin gene-related peptide (CGRP) plays a major role in the initiation of a cluster headache attack, possibly involving the ATP-sensitive potassium channels. The current study aims to determine whether the opening of ATP-sensitive potassium channels triggers cluster headache attacks in patients with cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* Cluster headache patients meeting ICHD-3 criteria for episodic and chronic cluster headache of either sex. Patients were defined as having episodic cluster headache in the active phase when they had usual attacks within the last 30 days, episodic cluster headache in the remission phase when they were attack-free for at least 30 days, or chronic cluster headache when they had not had more than 30 consecutively attack-free days over the last 12 months or longer.
* Weight between 50 and 100 kg.
* All preventive medications, except steroid treatments or greater occipital nerve blockade within 30 days, were allowed with stable dosing.
* Negative urinary HCG at baseline.

Exclusion Criteria:

* Primary headache types except above.
* Secondary headache disorders, according to ICHD-3.
* Headache at baseline.
* Anamnestic information or clinical signs of (at inclusion date) hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 50 mmHg)
* Known severe or treatment-requiring cardiovascular disease including cerebrovascular disease.
* Anamnestic or clinical evidence of mental disorder or substance abuse.
* Anamnestic or clinical evidence of any disease considered by the investigating physician to be relevant to participation in the study.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of cluster headache attacks | Change from baseline at 90 minutes after drug administration
  Experimentally induced cluster headache attacks must fulfill either:
  1. Headache described as mimicking the patient's usual cluster headache attack (with or without cephalic autonomic symptom).
  2. Headache fulfilling criteria A and B for cluster headache according to International Classification of Headache Disorders criteria:
  A. Severe unilateral pain lasting 15 to 180 minutes.
  B. Either or both of the following:
  * At least 1 cephalic autonomic symptom ipsilateral to the headache.
  * A sense of restlessness or agitation.

SECONDARY OUTCOMES:
Occurrence of headache | Change from baseline at 90 minutes after drug administration
  Yes/no questions.
Change of headache intensity scores | Change from baseline at 90 minutes after drug administration
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no headache; 1 is a very mild headache, including a feeling of pressing or throbbing; 5 is a moderate headache; 10 is the worst imaginable headache.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Khazali HM, Deligianni CI, Pellesi L, Al-Karagholi MA, Ashina H, Chaudhry BA, Petersen AS, Jensen RH, Amin FM, Ashina M. Induction of cluster headache after opening of adenosine triphosphate-sensitive potassium channels: a randomized clinical trial. Pain. 2024 Jun 1;165(6):1289-1303. doi: 10.1097/j.pain.0000000000003130. Epub 2023 Dec 19. PMID 38127692